MBARARA UNIVERSITY OF SCIENCE AND TECHNOLOGY

RESEARCH ETHICS COMMITTEE

P.O. Box 1410, Mbarara, Uganda

Tel. 256-4854-33795 Fax: 256 4854 20782

Email: irc@must.ac.ug mustirb@gmail.com

Web site: www.must.ac.ug









## INFORMED CONSENT FORM: RANDOMISED CONTROLLED TRIAL

This document outlines the research study and expectations for potential participants. It should be written in layman terms and typed on MUST-IRC letterhead. The wording should be directed to the potential participant NOT to IRC. If a technical term must be used, define it the first time it is used. Also, any abbreviation should be spelled out the first time it is used.

NB: All the sections of this document must be completed without any editing or deletions

Please use a typing font that is easily distinguishable from the questions of the form

Study Title: It should be the same as on all other documents related to the study

AFFECTING THE EPIDEMIOLOGY OF HIV IN UGANDA THROUGH OLDER ADOLESCENTS

Principal Investigator(s):

Emmanuel Kyagaba, Principal Investigator, Mbarara University of Science and Technology and Internet Solutions for Kids, Uganda Michele Ybarra, Ph.D., Principal Investigator and President, Center for Innovative Public Health Research (CiPHR)

## INTRODUCTION

HIV continues to be a significant public health challenge in Uganda.

## What you should know about this study:

- You are being asked to join a research study.
- This consent form explains the research study and your part in the study
- Please listen to it carefully and take as much time as you need to decide
- You are a volunteer. You can choose not to take part. And if you join, you may quit at any time. There will be no penalty if you decide to quit the study.

**Purpose of the research project:** Include a statement that the study involves research, estimated number of participants, an explanation of the purpose(s) of the research procedure and the expected duration of the subject's participation.

**Background/ Purpose** 

We are developing a sexual health and HIV prevention program for young adults in Uganda. The program will be sent to young people through text messages. This research study is

| Leave blank for IRC office only: | IRC OFFICE USE ONLY: |
|----------------------------------|--------------------------------------|
| | APPROVAL DATE: |
| MUST-IRC Stamp: | APPROVED CONSENT IRB VERSION NUMBER: |
| • | PI NAME: |
| | IRB NO: |

Michele Ybarra, MPH, PhD

Version Not Yet Approved by CIRBI

Page **1** of **4**